CLINICAL TRIAL: NCT00942032
Title: Clinical Experience With the Hindfoot Arthrodesis Nail (HAN) for the Surgical Treatment of Ankle and Hindfoot Pathologies. A Retrospective Case Series.
Brief Title: Clinical Experience With the Hindfoot Arthrodesis Nail for the Surgical Treatment of Ankle and Hindfoot Pathologies
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: Synthes Inc. (Industry)
Responsible Party: Andrew K. Sands, MD, St. Vincent's Hospital, Foot and Ankle Surgery
Organization: AO Innovation Translation Center (Other)
Other Study IDs: HAN-09
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Hindfoot Arthrodesis; Hindfoot Pathologies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this observational study is to collect and evaluate the current clinical experience gained from the Hindfoot Arthrodesis Nail (HAN) for ankle and hindfoot fusions.

DETAILED DESCRIPTION:
The HAN (Synthes) is a newly designed, titanium nail for trans-calcaneal, retrograde hindfoot fusion. The lateral bend allows an entry site in the center of the lateral column of the calcaneus, thus minimizing the risk of iatrogenic injury of the plantar neurovascular bundle.

ELIGIBILITY:
Inclusion Criteria:

* HAN fusion procedure ≥ 12 months before entering the study.
* Written or oral informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients will be identified from the study sites' medical records, information systems, and OR logs. The responsible local investigator or co-investigator at each study site will approach patients by letter or phone, and inquire about their interest in participating in this study.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2009-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The aim of this observational study is to collect and evaluate the current clinical experience gained from the Hindfoot Arthrodesis Nail (HAN) for ankle and hindfoot fusions. | More than 1 year

SECONDARY OUTCOMES:
Technical and surgical details Patient-centered endpoints (e.g., function as assessed by AAOS Foot and Ankle Outcomes Questionnaire (AAOS-FAOQ) score and the SF-36 Health Survey) | More than 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Beate P. Hanson, MD, Study Director — Ao Clinical Investigation and Documentation, Davos, Switzerland; Andrew K. Sands, MD, Principal Investigator — St. Vincent's Hospital, Foot and Ankle Surgery
Locations (7):
- United States (3):
  - Eisenhower Medical Center, Rancho Mirage, California
  - Medical University of South Carolina, Charleston, South Carolina
  - Harborview Medical Center, Seattle, Washington
- Centre Hospitalier Universitaire d'Angers, Angers, France
- Germany (2):
  - Charité Berlin, Campus Virchow Klinikum, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
- Stockholms Fotkirurgklinik Sophiahemmet, Stockholm, Sweden